CLINICAL TRIAL: NCT00784459
Title: Costimulation Inhibition in Asthma
Brief Title: The Effect of Inhibition of B7-mediated Costimulation on Allergic Airway Inflammation in Mild Atopic Asthmatics
Acronym: CIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jonathan Green, MD, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 08-0405
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2013-12

CONDITIONS: Atopic Asthma
Keywords: Asthma; Allergy
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with Abatacept (Experimental): Administration of Abatacept intravenously 10 mg/kg every 2 weeks for 3 doses, followed by every 4 weeks for 2 doses.
  Interventions: Drug: abatacept
- Placebo (Placebo Comparator): Administration of placebo (normal saline) intravenously 10 mg/kg every 2 weeks for 3 doses, followed by every 4 weeks for 2 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: abatacept — Treatment with abatacept, 10 mg/kg IV, for 5 doses.
  Other Names: Orencia; CTLA4Ig
  Arms: Treatment with Abatacept
Drug: Placebo — Treatment with Placebo, IV
  Arms: Placebo

SUMMARY:
This study is designed to determine if treatment with abatacept is effective in decreasing allergic airway inflammation in mild, atopic asthmatics. Subjects will be recruited from the greater St Louis Metropolitan area. Eligible individuals will undergo a titrated skin prick test. Following baseline evaluation, fiberoptic bronchoscopy with segmental allergen challenge (SAC) will be performed. The subjects will be randomized to either placebo or abatacept. After 12 weeks of study drug, the subjects will undergo repeat SAC. The primary endpoint will be to determine if treatment with abatacept results in a 50% or greater decrease in the percentage of eosinophils recovered in the bronchoalveolar lavage (BAL) fluid following SAC as compared to placebo control. Secondary endpoints include measures of airway obstruction and hyperreactivity, airway inflammation and symptoms as well as determination of the safety of abatacept administration in this subject population.

DETAILED DESCRIPTION:
please see summary

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. 18 - 50 years of age;
2. Previously documented physician-diagnosis of asthma consistent with NAEPP guidelines, with alternative diagnoses (eg, chronic obstructive pulmonary disease) ruled out;
3. Forced expiratory volume in one second (FEV1) ≥ 70% of predicted value at screening and at first SAC visit;
4. Positive methacholine inhalation challenge test of (PC20) ≤ 8 mg/mL within 6 months or at screening visit;
5. History of atopic symptoms by subject self-report (allergic rhinitis, conjunctivitis, or eczema);
6. A positive skin prick or intradermal test to cat allergen extract, short ragweed allergen extract, or dust mite allergen extracts at screening visit. A positive skin test is defined as induration of skin test wheal being ≥ 2 mm greater in diameter than saline control skin wheal;
7. After the baseline SAC (V3), subject should demonstrate at least a 50% increase in the percentage of eosinophils (compared to pre-allergen saline) and at least 10% eosinophils in post allergen lavage.
8. Stable asthma as reflected by no significant changes in controller asthma medications, no acute asthma exacerbations requiring oral corticosteroids, hospitalizations, emergency room visits, or unscheduled health care provider visits for asthma for at least 4 weeks prior to screening and up through the time of the first dose of study drug;
9. No history of intubation for asthma;
10. Sexually active women of childbearing potential must use an effective method of birth control during the entire course of the study and for 10 weeks after the final dose of the study drug, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential (WOCBP) will be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. All WOCBP MUST have a negative pregnancy test on the day of drug administration prior to receiving each dose. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study. In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
11. Ability to give informed consent (adults must be able to consent for themselves and be literate) and to comply with study procedures.

Exclusion Criteria:

Patients must have none of the following:

1. Lung disease other than allergic asthma (eg, chronic bronchitis, COPD);
2. Use of chronic oral corticosteroids or inhaled corticosteroids at doses > 440 μg/da fluticasone or equivalent within four weeks prior to screening visit
3. Concurrent diseases, finding on physical examination, or screening laboratory studies that, in the investigator's opinion, would interfere with participation in the study or that might put the participant at risk by participating;
4. Upper or lower respiratory tract infections within 4 weeks before screening;
5. No febrile illness (>38.0o C or 100.4oF) within 24 hours at screening and through the time of the study drug administration on Study Day 0;
6. Current use of any β-adrenergic antagonist (eg, propranolol)
7. Use of long acting beta-agonists (LABA) or long acting muscarinic antagonists (LAMA) within 2 weeks of screening visit.
8. Use of theophylline preparations.
9. Current allergy immunotherapy within 3 months of screening.
10. Use of systemic immunosuppressive drugs including systemic corticosteroids ,within the 4 weeks prior to screening up through administration of study drug;
11. Use of any TNFα inhibitor within 12 weeks of administration of study drug.
12. Participation in an intervention research study within past 4 weeks or receipt of any investigational drug or biologic(s) within 5 half-lives of the agent prior to the first dose of study drug and through Study Day 154;
13. Evidence of infection with hepatitis B or C virus, or human immunodeficiency virus-1 or 2 (HIV-1 or HIV-2), or active infection with hepatitis A;
14. History of cancer other than basal cell carcinoma or cervical carcinoma-in-situ that has been treated and cured by conization or other techniques.
15. History of primary immunodeficiency;
16. History of use of tobacco products of more than one cigarette per month or equivalent within 1 year prior to screening or history of smoking of greater than or equal to 10 pack-years;
17. History of a positive PPD;
18. History of allergic reaction to abatacept or any of the components of the study drug.
19. Pregnancy, women that are breast feeding, or that have an intention to become pregnant or breast feed during the time frame of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Green, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Parulekar AD, Boomer JS, Patterson BM, Yin-Declue H, Deppong CM, Wilson BS, Jarjour NN, Castro M, Green JM. A randomized controlled trial to evaluate inhibition of T-cell costimulation in allergen-induced airway inflammation. Am J Respir Crit Care Med. 2013 Mar 1;187(5):494-501. doi: 10.1164/rccm.201207-1205OC. Epub 2013 Jan 4. PMID 23292882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited from asthma patient subject registry
Groups:
- Placebo: Placebo : Treatment with Placebo, IV
- Treatment With Abatacept: abatacept : Treatment with abatacept, 10 mg/kg IV, for 5 doses.
Period: Overall Study
Arm/Group | Placebo | Treatment With Abatacept
Started | 11 | 13
Completed | 11 | 11
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment With Abatacept | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7.8) | 35 (9.8) | 31 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Baseline Percentage of Eosinophils Recovered in the BAL Prior to Segmental Allergen Challenge
Description: collected prior to randomization to abatacept or placebo
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Placebo | Treatment With Abatacept
Number analyzed (Participants) | 11 | 13
percentage of cells | 42 (30) | 19 (15)

2. Primary Outcome: Percentage of Eosinophils Recovered Following Segmental Allergen Challenge Following 3 Months of Placebo or Abatacept
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Placebo | Treatment With Abatacept
Number analyzed (Participants) | 11 | 11
percentage of cells | 44 (28) | 17 (17)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | Treatment With Abatacept
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days